

NHS
South London
and Maudsley
NHS Foundation Trust

Participant Identification Number: \_\_\_\_ Version 2.0

05/05/2018

## **CONSENT FORM**

Study Title: Can imagination change upsetting memories of trauma?

| 1. | | | sheet dated 05/05/2018 (version 2.0) uestions and had them answered in | Please<br>initial<br>boxes |
|---|---|---|---|---|
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I am willing for researchers to inform my clinical team that I am taking part in the project and provide information relevant to my care while I am taking part. I understand that this information will be added into my electronic notes. | | | |
| 4. | I allow the project team to access my clinical notes for information relevant to the project. This access will remain for the full time I am participating in the project. However, if I tell the team I do not want them to access my clinical information anymore, then they will stop. | | | |
| 5. | I understand that information relating to me taking part in this project will be anonymized (i.e. it will not contain my name) and stored on electronic database for up to 7 years. | | | |
| 6. | I know what to do if I have any concerns or want to make a complaint about any individual (e.g. the research therapist) or the project | | | |
| 7. | In order to check the quality of the project, I am willing for the meetings I have as part of the project to be audio recorded [this is optional] | | | |
| 8. | I give consent for quotations to be taken from the audio recordings for use in future teaching materials and publications. I understand that these quotations will be anonymous [this is optional]. | | | |
| 9. | I understand that if I am no longer able to provide informed consent during my involvement with the project, then my involvement will end at that point. I understand that the data collected before this point will still be used. | | | |
| 10. | I agree to take part in the above project. | | | |
| Name of Participant | | Signature | Date | |
| Name of person taking consent (if different from researcher) | | Signature | Date | |
| Researcher | | Signature | Date | |

<sup>\*1</sup> copy for participant; 1 copy for researcher site file; 1 copy for medical notes.